Official Study Title: Study of CPX-351 (VYXEOS) in Individuals < 22 Years With Secondary

Myeloid Neoplasms

CTG Number: NCT05656248

**Document Date:** 06/03/2025

# A PROSPECTIVE, SINGLE SITE, SINGLE-ARM PILOT STUDY OF CPX-351 (VYXEOS) IN INDIVIDUALS < 22 YEARS WITH SECONDARY MYELOID NEOPLASMS

**Note**: When we say "you" in this informed consent document, we mean "you or your child." When we talk about research, it can be called a clinical trial, research study (study), or research protocol.



## **Key Information**



To start, we highlight here the risks, benefits and study requirements that we think you should know before deciding if you want to take part in this research study. If you're still interested, we'll then get into more details.

A. Why are you being asked to voluntarily take part in this study?

You are being asked to take part in a research study because you have been diagnosed with a secondary myeloid neoplasm (leukemia, myelodysplastic syndrome, cancer) that was caused by previous cancer therapy you received or from a previous blood disease or syndrome. Secondary myeloid neoplasms are also called "SMNs".

B. What is the usual approach to your type of leukemia?

Many different treatment programs have been used for children with secondary myeloid neoplasms (SMNs). There is no standard therapy for SMNs, but most patients would have some type of chemotherapy followed by a bone marrow or stem cell transplant, if possible. You have a choice between other treatments for your SMN and this research study.

C. Why is this study being done?

The purpose of this study is to learn the effects (good and bad) of treatment with an investigational drug, CPX-351 (Vyxeos®) in patients with SMNs.

D. What will happen if you decide to take part in this study?

You will receive up to two cycles of chemotherapy with a drug called CPX-351.

E. What are the research risks and benefits of taking part in this study?

The most common side effects of CPX-351 are bruising and bleeding, low red blood cells (anemia), fever, chills, cough, shortness of breath, decreased appetite, infections, headache, mouth sores, nausea, vomiting, diarrhea, belly pain, constipation, muscle pain, skin rash, swelling, tiredness, difficulty sleeping and low blood pressure. Other side effects are listed in the "What are the risks and benefits of this study" section later in this consent.

The possible benefit is that the treatment on this study may cause your cancer to stop growing for a period of time or go into remission. It may also lessen the symptoms, such as pain, that are caused by the cancer or enable additional therapies, such as transplant.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 F. How many people will take part in this study?

Up to 25 children and young adults will take part in this study at St. Jude.

G. What are your options?

If you decide not to take part in this study, you have choices. For example:

- you may choose to receive other chemotherapy, not part of a research study
- you may choose to take part in a different study if one is available
- · or you could decide not to be treated

If you are still interested in taking part in this research study, CPXSMN, more detail is provided below in the following pages.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital IRB NUMBER: 22-1021

# Study Contact Details and Further Information

You are encouraged to ask any questions you wish, before, during or after your treatment. If you have any questions about the study, please speak to your doctor, who will be able to provide you with the up-to-date information about the drugs and procedures involved. If there is anything that you do not understand, or if you have any other questions, please contact any of the people below.

| Who to talk to for | You can contact | <u>At</u> |
|---|---|---|
| <ul> <li>Any new or unexpected symptoms, side effects or discomforts</li> <li>General study questions</li> <li>Research related injuries</li> <li>Any research concerns or complaints</li> <li>Any medical or surgical treatments done outside of St. Jude such as with your local doctor or another hospital during this study</li> </ul> | Raul Ribeiro, MD or your St. Jude<br>Doctor<br>262 Danny Thomas Place<br>Memphis, TN 38105 | 901-595-3300<br>(Main Hospital<br>Number) |
| Your rights as a research participant Any research concerns or complaints | Institutional Review Board (IRB)/Research Participant Advocate IRB is a group of scientists and community members who make sure research meets legal and ethical standards Research Participant Advocates are individuals who are not part of the research study team and are available to you to discuss problems, concerns and questions. The Advocate can help you obtain information and can relay any input you may have concerning the research to the research study team and the IRB. | or |

#### **Table of Contents**

| 40. | 1. | Why are you being asked to voluntarily take part in this research study? | 5 |
|---|---|---|---|
| *** | 2. | Who is sponsoring this study? | 5 |
| <b>@</b> | 3. | What is the purpose of the Study? | 5 |
| E | 4. | What will be done in this study? | 6 |
| $\overline{\Psi}$ | 5. | What are the risks and benefits of being part of this study? | 9 |
| <b>†</b> } | 6. | What are the reproductive risks of being part of this study? | 13 |
| 0 | 7. | Can you stop taking part in this study? | 13 |
| \$ | 8. | What are your other options, and can you have other treatments while taking part in this study? | 18 |
| \$ | 9. | How much will it cost to take part in this study? | 14 |
| <u></u> | 10. | Will I be paid for my time or expenses? | 15 |
| • | 11. | What if there is a problem? | 15 |
| 7 | 12. | How will new findings related to your participation this study be shared with you? | 15 |
| | 13. | How will you find out results of this study? | 15 |
| ₹ | 14. | Will any genetic testing be done, and what are the risks of genetic testing? | 16 |
| | 15. | What about identifiable private information and identifiable biospecimens? | 17 |
| Ø | 16. | What about permission to use your data/information (HIPAA), privacy, and confidentiality? | 19 |
| | 17. | Signature Pages | 23 |



# 1. Why are you being asked to voluntarily take part in this research study?

You are being asked to take part in a research study because you have been diagnosed with a secondary myeloid neoplasm (leukemia, myelodysplastic syndrome, cancer) that was caused by previous cancer therapy you received or from a previous blood disease or syndrome. A myeloid neoplasm is a type of disease in which the bone marrow makes too many or too few red blood cells, platelets, or certain white blood cells. These types of diseases are also called secondary myeloid neoplasms or SMNs.

This consent form gives you information about the study that will be discussed with you. Please take your time making a decision and feel free to discuss it with your friends, family and St. Jude staff. Before agreeing to take part in this research study, it is important that you read this consent form that describes the study. After you understand the study, and if you agree to take part, you will be asked to sign this consent form. You will be given a signed copy to keep.

Your participation in this research study is entirely voluntary. You may refuse to participate or stop your participation at any time.



## 2. Who is sponsoring this study?

This study is being sponsored by St. Jude Children's Research Hospital. The drug manufacturer, Jazz Pharmaceuticals, is supplying CPX-351 at no charge to St. Jude for this study.

The principal investigator (researcher) in charge of this study is Dr. Raul Ribeiro. He may be reached by phone at present the study is Dr. Raul Ribeiro. He may be reached by the study is Dr. Raul Ri



## 3. What is the purpose of this study?

The purpose of this study is to learn the effects (good and bad) of treatment with an investigational drug, CPX-351 in patients with SMNs. With this research study, we plan to meet the following goals:

- Find out if CPX-351 is an effective treatment for SMNs
- Learn more about the side effects of this treatment
- Learn more about the body reacts to CPX-351
- · Learn more about the biology and genetics of patients with SMNs

Up to 25 participants will take part at St. Jude.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital IRB NUMBER: 22-1021



## 4. What will be done in this study?

#### Before you start treatment

You will need to have the following exams, tests or procedures to find out if you can be in the study. These exams, tests or procedures are part of regular cancer care and may be done even if you do not join the study. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

- History and physical exam
- Blood counts and chemistry to test the function of your bone marrow, liver and kidneys.
   About a teaspoon of blood will be obtained.
- Pregnancy test (if you are a female who could have children)
- . Bone marrow aspirate and biopsy to check the status of your leukemia
- Lumbar puncture (spinal tap) to check the fluid around your spine and brain for leukemia cells
- Electrocardiogram (ECG) and Echocardiogram (ECHO) to test the function of your heart

Because of the possible risk of heart damage with CPX-351, you cannot take part in this study if you have already received too much doxorubicin (or similar drugs known to cause heart damage) in the past. If you have not received doxorubicin in the past, the equivalent dose of doxorubicin will be calculated based on the drug (daunomycin, idarubicin, epirubicin and mitoxantrone) you did receive during your prior therapy to determine whether or not you are eligible for this research study.

If the test results show that you do not meet the study eligibility, you cannot start the study treatment and your study doctor will talk to you about other treatment options.

#### During the study

If the exams, tests and procedures show that you can be in the study, and you choose to take part, you can start treatment.

One cycle of treatment is shown below.

| Drug | How the drug will be given | No. of doses | Days |
|---|---|---|---|
| CPX-351 (cycle 1) | Into the vein over about 90 minutes (IV) | 3 | Days 1, 3 and 5 |
| CPX-351 (cycle 2) | Into the vein over about 90 minutes (IV) | 2 | Days 1 and 3 |
| Intrathecal chemotherapy (methotrexate, | Into the fluid surrounding the brain and spinal cord (IT) | 1 | Day 1 of each cycle |

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025

| Drug | How the drug will be given | No. of doses | Days |
|---|---|---|---|
| cytarabine and hydrocortisone) | | | |

You can receive up to 2 cycles of this treatment (about 2 months). After that, you will proceed either to allogeneic hematopoietic stem cell transplant (HSCT) or other therapies as your doctor recommends. If you attain remission (no signs of disease) after the first course of CPX-351, and HSCT transplant can occur within 3 to 4 weeks from the start of the first course, you can proceed to HSCT without receiving the second course of CPX-351.

## Other therapies

If you are scheduled to have an allogeneic transplant but there will be a delay in timing, your study doctor may decide to administer an additional cycle of CPX-351 or other chemotherapy drugs. Your study doctor will discuss this with you and obtain another informed consent if drugs other than CPX-351 is necessary.

Intrathecal (IT) chemotherapy to prevent or treat leukemia in the spinal fluid

You may be familiar with spinal taps if they were done during the initial treatment of your primary cancer. Whether you decide to take part in this study or not, you will need additional spinal taps to give medicines that are necessary to prevent the leukemia from spreading to your spinal fluid, or to treat the spinal fluid if leukemia cells are present.

All patients will get one IT chemotherapy treatment with methotrexate, cytarabine and hydrocortisone before or right after starting the first cycle. Additional doses of IT chemotherapy will depend on whether or not you have leukemia cells in your spinal fluid and how many relapses of leukemia you have had before starting this study. You will also receive a vitamin supplement called leucovorin, which will help prevent or lessen side effects of the IT chemotherapy.

You will get some form of sedation or anesthesia (medicine to make you sleep) during this procedure. Spinal taps are painful and may cause headaches. The skin at the site of needle insertion is usually numbed with an anesthetic cream or lidocaine before the procedure is performed. About 1 teaspoon of spinal fluid will be withdrawn before injecting the chemotherapy.

#### Recovery and leukemia evaluation after treatment

You may need to be in the hospital for the administration of this treatment. It will take 2-3 or more weeks for your blood counts to fully recover from this treatment. After three weeks from the first day of treatment, a bone marrow exam will be done to evaluate the status of your leukemia (measurement of residual disease or MRD).

#### Standard of care tests and procedures during treatment

During treatment on this study, you will have the following tests and procedures that are part of standard of care for leukemia:

Physical exam and vital signs will be done regularly during treatment

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital IRB NUMBER: 22-1021

- Blood tests to check your blood counts and blood chemistry will be done regularly during treatment. About a teaspoon of blood will be obtained.
- Lumbar puncture (spinal tap) to check the fluid around your spine and brain for leukemia cells
- Electrocardiogram (ECG) and Echocardiogram (ECHO) to test the function of your heart
- Pregnancy test (if you are a female who could have children)
- Bone marrow exams before and at the end of treatment to evaluate comprehensive leukemia genomics and the amount of residual leukemia in the bone marrow. The measurement of residual disease (MRD) indicates the your leukemia's response to treatment

### Required research studies during this study

The following tests will be done because you are part of this study. If you were not in the study you would probably not have these tests. The information learned would not change the way you are treated. With the exception of the genetic studies mentioned below, the results of these tests will not be given to you. You and your insurance company will not be charged for the costs of the required research study tests listed below.

## Pharmacogenomics

If you will receive a HSCT after treatment on this study is completed, a blood sample will be collected for pharmacogenomic research studies. About 1 teaspoon of blood will be collected for this research study. This type of research is done to study how a person's genes may affect the way he or she responds to treatment.

#### Genomic studies

You have previously signed a clinical genomics consent that gives more detail about genetic testing. Both leukemia and normal cells will be tested. These results will be provided to your study doctor. They will only receive results that show specific genetic changes that may affect how you respond to the study drugs.

Your tumor and non-tumor DNA will be sequenced. We will use your bone marrow (about 2 teaspoons) and your blood (about 1 teaspoon) collected at the same time you are having clinical procedures. Researchers are looking for changes in DNA that may be related to the development of leukemia, or that may explain why some patients might respond to certain treatments better than other patients. Some of the changes may be present in every cell of the body, including leukemia cells and normal cells (germline mutations), while other changes may only be present in the leukemia cells (somatic mutations).

You will also be asked to sign our TBANK consent, which allows the St. Jude "biorepository" to store your blood and tissue, including your DNA, for the research objectives of this study and, beyond this study, for other future research. The TBANK consent also gives more detail on how your genetic results may be used and shared in the future.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital

IRB NUMBER: 22-1021



## 5. What are the risks and benefits of taking part in this study?

#### a. Risks

If you choose to take part in this study, there is a risk that you may:

- Lose time at school, work or home and spend more time in the hospital or doctor's office than usual
- Be asked sensitive or private questions which you normally do not discuss

The chemotherapy drug used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and bone marrow (blood). The study doctor will be testing your blood and will let you know if changes occur that may affect your health. There is also a risk that you could have side effects.

Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- · Some side effects may interfere with your ability to have children.
- · Some side effects may be serious and may even result in death.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.

#### Infection

There is a serious risk of developing an infection while being treated on this research study, including serious infections that may require hospitalization. To reduce the risk of developing an infection, you will be required to take antibiotics and antifungal medication. You may be required to be in the hospital for most of the treatment so that your doctors and nurses can monitor you very carefully for any signs or symptoms of infection.

If you experience any of the following signs or symptoms while you are being treated on this research study, it is very important to call your doctor or nurse right away.

- Fever
- Pain (earache, sore throat, headache, pain with urination or having a stool)
- · Redness, swelling, pain, or pus at the site of your central catheter

Risks of the study

Harmful reactions or side effects may occur in patients taking part in research studies. Some of these will be due to the patient's disease or prior treatment and some may be due to the drug being studied. Everyone taking part in the study will be watched carefully for any side effects. However, doctors don't know all the side effects that may happen. In general, side effects can range from mild to serious. Your health care team may give you medicines to help lessen side effects. Many side effects go away soon after you stop treatment. Although numerous measures are established to protect your health, it is possible that in some cases, side effects can be serious, long lasting, or may never go away.

Patients with leukemia may have a risk of death due to their underlying cancer or as a complication of their cancer treatment. Side effects related to this treatment will be closely monitored.

#### Unknown risks

The drug combination is experimental and still being tested. There may be other risks, including death, which are not known now.

Possible side effects of CPX-351 include:

## COMMON, SOME MAY BE SERIOUS

In 100 people receiving CPX-351, more than 20 and up to 100 may have:

- · Bruising, bleeding
- Anemia which may require blood transfusion
- Fever, chills
- Cough, shortness of breath
- Decreased appetite
- Infection, especially when white blood count is low
- Headache
- Mouth sores

- Nausea, vomiting, diarrhea, pain in the belly, constipation
- Muscle pain
- Rash
- Swelling of the body
- Tiredness
- Difficulty sleeping
- Low blood pressure which may cause feeling faint

## OCCASIONAL, SOME MAY BE SERIOUS In 100 people receiving CPX-351, from 4 to 20 may have:

- Dizziness
- Heartburn
- Worry, sudden confusion
- Itching
- Fluid around the lungs which may cause shortness of breath
- High blood pressure which may cause headaches, dizziness, blurred vision
- Abnormal heartbeat
- · Increased sweating or night sweats
- Kidney damage which may require dialysis
- Damage to the lungs which may cause shortness of breath
- Chest pain
- Problems with vision
- Heart failure which may cause shortness of breath, swelling of ankles, and tiredness

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025

IRB NUMBER: 22-1021

#### RARE, AND SERIOUS

In 100 people receiving CPX-351, 3 or fewer may have:

- · Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- · Redness, pain or peeling of palms and soles
- Increased blood copper levels

In addition to the risks described above, there may be unknown risks, or risks that we did not anticipate, associated with being in this study.

Possible side effects of INTRATHECAL TREATMENT (spinal injection of methotrexate, cytarabine and hydrocortisone, or cytarabine alone) include:

#### COMMON, SOME MAY BE SERIOUS

- Nausea and/or vomiting
- Fever

Headache

#### OCCASIONAL, SOME MAY BE SERIOUS

- Swelling of the brain, which may cause stiff
   Difficulty learning neck, sensitivity to light, headache, vomiting
- Major change in thinking patterns
- Confusion
- Tiredness
- Seizure

#### RARE, AND SERIOUS

- Rash
- Bleeding in the brain
- Paralysis, weakness

- Dizziness
- Damage to the brain, which may cause changes in thinking, blindness
- Infection

Possible side effects of LEUCOVORIN CALCIUM include:

#### COMMON, SOME MAY BE SERIOUS

In 100 people receiving leucovorin, more than 20 may have:

- Diarrhea, nausea, vomiting
- Sores in mouth, which may cause
  - difficulty swallowing

Tiredness

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving leucovorin, from 4 to 20 may have:

· Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat

#### RARE, AND SERIOUS

In 100 people receiving leucovorin, 3 or fewer may have:

None

Leucovorin is a vitamin supplement that is given to decrease the side effects of methotrexate.

Some drugs or supplements may interact with your treatment plan. Talk to your doctor, pharmacist, or study team before starting any new prescription or over-the-counter drugs, herbals, or supplements and before making a significant change in your diet. Supplements

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital

IRB NUMBER: 22-1021

may come in many forms, such as teas, drinks, juices, liquids, drops, capsules, pills, or dried herbs. All forms should be avoided.

If your red blood cell count is low, the cells that carry oxygen around the body, you may feel tired. If your red blood cell count drops very low you may need a blood transfusion.

If you have a decrease in the white blood cell count, the cells that fight infection, you may be more likely to get an infection, including a serious infection that spreads through the blood stream (sepsis). If this happens, you will have to come to the hospital to be treated with antibiotics. If your white blood cell count is very low and you get a fever, you may have to come to the hospital to get treated with antibiotics.

If you have a low platelet count, particles in the blood that help with clotting, you may have easy bruising or bleeding. If the count is very low or there is bleeding, you might need platelet transfusions to help stop the bleeding.

### Loss of privacy

Very rarely, personal information from your records could be given out by accident. This might make you upset, embarrass you, or affect your ability to get insurance. Additional privacy and other risks from genomic testing are discussed in the clinical consent. To stop this from happening, we:

- Store records apart from names or other personal information
- Only allow members of the study team to see the records
- Store electronic data only on computers protected with a password and encryption software
- Report study results on the whole group and never identify one single person in any reports

#### b. Benefits

We hope that this study will help you personally, but we do not know if it will.

The potential benefits of treatment on this study include:

- May cause your cancer to stop growing for a period of time or go into remission.
- May lessen the symptoms, such as pain, that are caused by the cancer or enable you to receive additional therapies such as HSCT.

With any cancer treatment, sometimes treatment does not make the cancer go away. Sometimes treatment makes the cancer go away for a while but the cancer comes back later.

Information learned from this study may benefit other patients in the future.

Revision 2.1 dated: 03-31-2025

Consent document date: 03-31-2025

St. Jude Children's Research Hospital

IRB NUMBER: 22-1021



6. What are the risks to pregnancy, to an unborn child, and to the ability to have children (fertility) when taking part in this study?

Females should not become pregnant and males should not father a baby while on this study because the drug(s) in this study can be bad for an unborn baby. If you or your partner can get pregnant, it is important for you to use birth control or not have sex while on this study and for 6 months after the last dose of CPX-351. Check with your study doctor about what kind of birth control methods to use and how long to use them. Some birth control methods might not be approved for use in this study. If you are a woman and become pregnant or suspect you are pregnant while taking part in this study, please inform your study doctor immediately. Females should not breastfeed a baby while on this study. Also check with your doctor about how long you should not breastfeed after you stop the study treatment.



## 7. Can you stop taking part in this study?

#### a. Can you change your mind about participating in this research study?

You may change your mind about taking part in this research study or stop at any time. The decision will not affect your care or your relationship with your doctor or St. Jude. If available, you may receive routine medical care at St. Jude Children's Research Hospital.

If you change your mind about participating in this study, samples or related information that have already been given to or used by researchers will not be returned or removed.

#### b. Can you be taken out of this study without your consent?

Your St. Jude doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest,
- If new information becomes available,
- If you do not follow the study rules,
- If the study is stopped by the sponsor, St. Jude

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital

IRB NUMBER: 22-1021



■ ■ 8. What are you other options and can you have other treatments while taking part in this study?

#### a. Other Treatment Options

If you decide not to take part in this study, you have choices. For example:

- you may choose to receive other chemotherapy, not part of a research study
- you may choose to take part in a different study, if one is available
- or you could decide not to be treated

#### b. Can you participate in other research studies at the same time?

Please check with your study doctor before thinking about taking part in any other research.

### c. Other medications, vitamins, and supplements

While in this study, you may not be able to take some or all of the medications or treatments you have been taking for your condition or for other reasons. It is important to tell your study doctor and the study staff about any treatments or medications you may be taking, including over-the-counter medications, vitamins or herbal remedies, acupuncture, or other alternative treatments.

Tell your study doctor about any changes to these during your participation in the research study. Your study doctor will explain to you which treatments or medications need to be stopped for the time you are involved in the research study.



## 9. How much will it cost you to take part in this study?

If you have health care coverage, we will bill your health care insurer for all standard of care services, tests, and procedures, as applicable. Billing your health care insurer impacts your annual deductible. This may affect your health care coverage to some extent if you go to another health care provider or institution in the future.

At St. Jude, you will not be responsible for or receive bills for co-pays, co-insurance, deductibles, or similar patient-liability amounts, or for the cost of medical care related to your disease or this study not covered by your health insurer. This includes research-only costs. Research-only tests and procedures will not be billed to you or your health care insurer.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025

IRB NUMBER: 22-1021

IRB APPROVAL DATE: 06/03/2025

St. Jude Children's Research Hospital



## 10. Will you be paid for your time or expenses while taking part in this study?

You will not be paid for your time or expenses.



## 11. What if there is a problem while taking part in this study?

If you are injured from being in this research study, please notify your St. Jude Doctor or the study doctor, Dr. Raul Ribeiro. St. Jude will offer you reasonable and necessary medical treatment for that injury. If you need more care than St. Jude can provide or if you prefer to seek treatment elsewhere, we will help you find medical care somewhere else. St. Jude may bill your insurance company or other third parties, if appropriate.

It is not the hospital's policy to provide payment for other types of costs, such as lost wages, disability, or discomfort if you are injured from being in this study. You are not giving up any of your rights by signing this consent form.



# 12. How will new findings related to your participation in this study be shared with you?

You will receive results from all the standard of care tests and procedures, including genetic testing. You will not receive results from the research studies, since they will not impact your care.

The researcher will tell you of any new information learned during your study participation which might cause you to change your mind about continuing the study.



## 13. How will you find out the results of this study?

St. Jude researchers share information with people in studies in many ways including:

- Articles on <u>www.stjude.org</u>
- In newsletters
- · In medical or scientific journals
- In the media
- A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> as required by the U.S. Law. This website will not include information that can identify you.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital

IRB NUMBER: 22-1021

At most the website will include a summary of the results. You can search this website at any time.

Published research results will only describe groups of people who took part in the study. Information that points out a single person will not be in research journals or other reports.



## 14. Will any genetic tests be done and what are the risks of genetic testing?

This study involves reading through all your genetic material to find certain changes that may explain information about you and/or your health condition (like how your health condition relates to other conditions, how certain drugs affect you or your health condition, etc.). The genetic material, or genes, are stored in your cells. The genetic material will be obtained from your sample (i.e., tumor, blood, skin, etc.). Information obtained from reading through your genes, as well as information about your health condition, will be entered into one or more scientific repositories or databases maintained by St. Jude Children's Research Hospital, the Federal Government, the European Genome-phenome Archive, or others.

#### Risks of Somatic Genetic/Genomic Testing

From the tumor testing alone, it may not be possible to tell if a genetic change is likely inherited or inheritable, or if it is only present in the tumor/cancer cells. To find out if a genetic change is inherited or able to be passed on to your children, your normal tissue sample would need to be tested. If you want to have your normal tissue tested, you should talk to your doctor to learn how this can be done.

It is possible that testing your tumor/cancer tissue will not help us better understand or find a cause of your disease or help us recommend a treatment. Most tests are not perfectly correct. There is also a chance that there could be an error in the testing or analysis.

After learning your results, you might feel anxious, upset or frustrated. Your doctor can discuss these concerns with you and arrange for needed follow-up, such as with the Genetics Service or other support services (social work, spiritual care, or psychology).

The genomic test report will be placed into your electronic medical record and may be seen by your other doctors and health care workers at St. Jude or other facilities that obtain your medical record with your permission or legal authority.

#### Risks of Germline Genetic/Genomic Testing

There is a chance that the genomic test results of your normal tissue will show that you have an inherited health condition, or a condition that can be passed down to any children you have. The condition discovered might show that you and possibly other family members are at risk of developing tumors or at risk of developing other health problems unrelated to cancer. It is also possible that testing your normal tissue sample will not find any genetic changes that will affect your current management or future health risks. Sometimes, genetic testing can find gene changes that we do not completely understand. This uncertainty may lead to anxiety or confusion.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital

IRB NUMBER: 22-1021

After learning your results, you might feel anxious, upset or frustrated. Your doctor will discuss these concerns with you and arrange for needed follow-up, such as with the Genetics Service or other support services (social work, spiritual care, or psychology).

When the genomic test report comes from a CLIA certified laboratory, the results will be placed into your electronic medical record and may be seen by your other doctors and health care workers at St. Jude or other facilities that obtain your medical record with your permission or legal authority.

Currently, the U.S. law known as the "Genetic Information Nondiscrimination Act" (GINA) prohibits discrimination based on genetic findings in some circumstances:

- a. GINA prohibits health care insurers from requesting or requiring genetic information of an individual or an individual's family members or using genetic information for decisions about health insurance coverage or rates, or to exclude preexisting conditions.
- b. In companies of 15 or more employees, GINA prohibits employment and employeerelated decisions from being made on the basis of genetic information of an individual or an individual's family members.

GINA protections do not apply to:

- a. the presence of disease or a health disorder,
- b. life insurance, long-term care insurance, or disability insurance. These insurance companies may consider this information in making insurance decisions affecting you,
- both health care plans and employment from companies employing fewer than 15 people, and
- d. people in the military.
- e. There are other health plans that GINA does not apply. Please ask your study doctor if you have any questions.



15. What about identifiable private information and identifiable biospecimens (blood, tissue, urine, cells, and any type of data and/or samples) obtained from you during the study?

If you choose to take part in this study, your data and/or specimens will be used to answer the research question(s) and to publish the findings of this study. Published research results will only describe groups of people who took part in the study. Information that points out a single person will not be in research journals or other reports. You will not own your research data and/or specimens. If researchers use your data and/or specimens to create a new product or idea, including those that may have commercial value, you will not benefit financially. There is no plan to share any money with you.

St. Jude's researchers and their collaborators will store the data and specimens collected in this study in electronic databases and other locations and will store specimens in the biorepository or other locations. They may use the data and/or specimens collected in this study for future research purposes and may share some of the data or specimens with others without seeking further consent from you. You may not receive results from that future research.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital

IRB NUMBER: 22-1021

Research Participant ID #: Research Participant Name:

CPXSMN Page 18 of 24

Sharing data and/or specimens is part of research. It may increase what can be learned from this study and future studies. Often data sharing is required as a condition of funding or for publishing study results. It is also needed to allow other researchers to validate study findings and to come up with new ideas.

Your data and/or specimens may be shared with government agencies, research collaborators, and other researchers and organizations conducting research that may not be related to this study. Your data may also be put in government or other databases/repositories as mentioned in the section above "Will any genetic tests be done and what are the risks of genetic testing?"

Future research using your samples and data is likely to include studies that look at genomic and genetic information to understand causes and cures for health conditions. Because science constantly advances, we do not yet know what other future uses of research data and/or specimens may include. There is no time-limit on sharing of information.

This future research may be unrelated to the current study and may include outside researchers and organizations from around the world. These organizations may include for-profit companies conducting medical research. We or others who distribute data or samples may be paid for data or samples, including yours. You will not receive payment if this happens.

St. Jude will do its best to protect and maintain your data and/or specimens in a safe way. One of the ways we protect your data and/or specimens is by limiting the uses of the information and the type of information that is shared, especially your personal information. This may occur through data sharing agreements and review by oversight groups within St Jude. Often the data and specimens may be coded to protect your identity before they are shared, and we will keep the key to the code in a secure way.

If data and/or specimens are used or shared with any information that may be likely to identify you, such as your name, address, or medical record number, further institutional review and approval would be required. In these cases, we will review whether additional consent from you is required.

Generally, if your data and/or specimens are used and shared without any personal identifiers or only with information that is less likely to identify you (such as the date of a procedure), further review and approval is not needed, and you will not be contacted.

By signing this consent form, you allow the drug manufacturer, Jazz Pharmaceuticals, to use study data and/or specimens for commercial purposes, and to use and share data and/or specimens from this study in the future for this and other studies. St. Jude may also use and share study data and/or specimens for patient care, academic uses, and publication, and when required by law. St. Jude and Jazz Pharmaceuticals will take precautions to remove any information that could identify you (like your name or medical record number) before sharing.

Data sharing could change over time and may continue after the study ends.

The use and sharing of your data and/or specimens is required for participation in this research study. The purpose of research is to learn and discover new information to make improvements to patient care and/or treatments. To make these improvements, research results must be shared with others. By agreeing to take part in research studies, you are agreeing for your information or data to be used and shared with others. If you are generally not comfortable with

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital

IRB NUMBER: 22-1021

the use and sharing of your data and/or specimens in future research as explained this consent, you should talk with your doctor before agreeing to take part in this study.



16. What about permission to use your data/information (HIPAA Privacy Rule), privacy and confidentiality?

#### Permission to Use Your Data/Information- HIPAA Privacy Rule and Privacy

The HIPAA Privacy Rule defines the situations in which PHI (protected health information) may be used or given to someone outside of the hospital to be used or released for research and other purposes. PHI includes information such as your name, MRN, date of birth, or other identifying information, including research information placed in your medical record.

To do this research, St. Jude Children's Research Hospital (St. Jude) will need to collect, use, and share your private health information. St. Jude is required by law to protect your health information. By signing this consent form, you give St. Jude permission to use and/or release (share) your private health information for this research. Those persons who receive your health information may not be required by Federal privacy laws (such as the Privacy Rule) to protect it and may share your information with others without your permission, if permitted by laws governing them.

If you sign this consent form, you give permission to all researchers and their staff involved in the study at St. Jude to use or release (share) your health information that identifies you for the research study described in this document.

The health information that we may use or release includes things learned from the procedures and treatments describes in this consent form, as well as all information from your medical record (which may include information such as HIV status, drug, alcohol, or STD treatment, genetic test results, or mental health condition and/or treatment, physical examinations, and lab tests). This may include, for example, all information in a medical record, results of physical examinations, medical history, lab tests, or certain health information indicating or relating to a particular condition.

If you sign this consent form, you give St. Jude permission to share your information for future research studies about disease or advancing science and for future unspecified research. You also give permission for us to place this information on databases as described below under Privacy and Confidentiality.

Information from research testing will be analyzed in a CLIA-certified (medical) laboratory or a research-only laboratory. By signing, you give St. Jude permission to put your research information obtained from a CLIA-certified laboratory into your medical record. Results from research-only laboratories will not be put into your medical record and will not generally be available to you or your doctor.

Any information placed in the medical record becomes a permanent part of your record, is kept indefinitely, It is protected like any other part of your medical record as described in the Notice of Privacy Practices. You have the right to see, copy, and ask for changes to your PHI that will be

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital IRB NUMBER: 22-1021

used or shared. However, research information may not be available until after the end of the study.

When you first registered at St. Jude, you received a copy of the St. Jude Notice of Privacy Practices. It tells how your PHI, including research information placed in your medical record, may be used or given to someone outside of St. Jude. You have the right to read the Notice of Privacy Practices before you sign this consent form. It may have changes since you first registered at St. Jude. You can find it at the bottom of every page on the St. Jude internet website: <a href="https://www.stjude.org">www.stjude.org</a>

The people who may view, request, receive, or use your private health information include St. Jude researchers and their staff, and other doctors, nurses, and staff members. Additionally, St. Jude may share your information with other people or groups of people. These include:

- Food and Drug Administration (FDA)
- Office of Human Research Protections (OHRP)
- National Institutes of Health (NIH)
- Other government agencies
- Your insurance company and other health benefits plan, including government coverage such as Medicaid
- Accrediting agencies like the Joint Commission and the College of American Pathologists
- St. Jude Children's Research Hospital Institutional Review Board (IRB)Other committees or people involved in overseeing research studies
- Others who have access to your medical record by authorization or law
- Jazz Pharmaceuticals (the drug manufacturer of CPX-351)

You do not have to sign this consent form which gives your permission, but if you do not, you may not receive research-related treatment.

Please note that you may change your mind and take back (revoke) this permission at any time. Even if you take back this permission, St. Jude Children's Research Hospital may still use or disclose health information they already have obtained about you as necessary to maintain the integrity or reliability of the current research. To take back this consent form/permission, you must write to:

| HIPAA Privacy Office | er |
|---------------------------------------|----|
| St. Jude Children's Research Hospital | |
| Memphis, TN | |

This permission does not have an expiration date.

#### Confidentiality

We will protect the confidentiality of your information to the extent reasonably possible.

Researchers and study staff are required by law to report suspected child abuse, threat of harm to self or others, and certain diseases that spread from person to person.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital IRB NUMBER: 22-1021

If you consent to take part in this study, information obtained from this study, as well as information about disease signs and symptoms, will be entered into one or more scientific databases maintained by St. Jude Children's Research Hospital and the Federal Government. The information will be held securely electronically at St. Jude Children's Research Hospital. Your name will not be passed on to anyone else outside the research team who is not involved in the study. You will be allocated a study number, which will be used as a code to identify you on all study forms. Any research-related information about you that leaves the hospital will have your name and address removed so that you cannot be recognized.

Research data obtained from this study from standard of care tests and procedures and research tests and procedures such as tumor and normal specimens and genetic data, are often shared with the research community using various databases, including those maintained by St. Jude, the federal government, and international collaborative databases. This is to advance scientific discovery, and to satisfy requirements of organizations that fund research, and journals that publish the results of research.

There are two types of databases used for sharing research data. One is a public, unrestricted access database and the other is a controlled access database. Each is described below.

#### Unrestricted access databases:

The information from research studies using your samples, genetic information, and some health information may be freely available in a public, unrestricted database that anyone can use. A public database could include information on hundreds of thousands of genetic variations in your DNA code, as well as your ethnic group and sex. Summary-level information about all participants included in a dataset, including you, but not genetic data for each individual, may be shared.

Some examples of information that may be shared includes how different genes are associated with different traits or diseases across the many participants in the dataset, or how often certain gene changes are seen across participants from many studies. However, the risk of anyone identifying you with this information is very low. This public information will not be labeled with your name or other information that could be used to easily identify you.

#### Controlled access databases:

Your individual genomic data and health information may be put in a controlled-access database. This means that only researchers who apply for and get permission to use the information for a specific research project will be able to access the information. Your genomic data and health information will not be labeled with your name or other information that could be used to easily identify you.

Researchers approved to access information in the database must agree to protect the information and not to try to identify you. Examples are the St Jude Cloud, which is run by St. Jude, the database of Genotypes and Phenotypes which is run by the Federal Government, and the European Genome-Phenome archive. These are databases available to researchers to use genomic information from tumor and non-tumor samples to study genetic changes in pediatric diseases.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025

cument date: 03-31-2025 IRB NUMBER: 22-1021 IRB APPROVAL DATE: 06/03/2025

St. Jude Children's Research Hospital



If you decide you would like to take part in this research study, please ask any questions you have, and read and sign this consent form. You will be given a copy of it to keep. A copy of this consent form will also be put in your patient notes, one will be put with the study records, and one may be sent to the Research Sponsor.

You can have more time to think this over if you are at all unsure.

Thank you for taking the time to read this informed consent document and to consider taking part in this study.

| Research Participant ID #:<br>Research Participant Name: | | | CPXSN<br>Page 23 of | |
|---|---|---|---|---|
| 17. Signatures | | | | |
| PARENT/GUARDIAN STATEMENT (Required this document or it was read to me. I questions have been answered. I give per | have been encoura | ged to ask qu | estions and all my | |
| | | | AM/F | РМ |
| Parent/Legal Guardian Signature | Date | Time | (circle one) | |
| ASSENT DISCUSSION (Required for part | icipants 7-13 years | old): | | |
| The research was explained to the min verbally agreed to take part in the stu | | e-appropriate | terms and the min | nor |
| Minor declined to take part in the study | . The minor decline | d for the follo | wing reason(s): | |
| ── An assent discussion was not initiated v | with the minor for th | e following re | ason(s): | |
| ☐ Minor is under 7 years of age. | | | | |
| Minor is incapacitated. | | | | |
| ☐ Minor refused to take part in the dis☐ Other | scussion. | | | |
| RESEARCH PARTICIPANT STATEMENT older): I have read this document or it was and all my questions were answered. I agr | read to me. I have | been encoura | aged to ask questic | |
| | | | AM/I | DM |
| Research Participant Signature | Date | | Time (circle or | |

IRB NUMBER: 22-1021

Research Participant ID #: Research Participant Name:

CPXSMN Page 24 of 24

| RESEARCHER/DESIGNEE STATEMENT his/her parent(s) or legal guardian(s). The encouraged to ask questions and all questithis form has been given to the participant | research participan<br>ions were answered | t and paren<br>d to their sa | t(s)/guar | dian(s) were |
|---|---|---|---|---|
| | | | | AM/PM |
| Researcher/Designee Signature | Date | | Time | (circle one) |
| Print Name | | | | |
| Interpreter (if needed) Signature | Date | Time | | AM/PM<br>(circle one) |
| RESEARCH PARTICIPANT ADVOCATE Sprocess. The research study, intervention/opresented to the research participant and/oquestions, and research team members an indicated that they: 1) understood the inforconsented/agreed to take part in the research | observation, risks, bor legal guardian(s)<br>nswered all their qua<br>mation presented; a | penefits, and<br>They were<br>estions. The | d alternat<br>encoura<br>participa | tives were<br>ged to ask |
| Research Participant Advocate | Date | _ | Time | AM/PM<br>(circle one) |
| Interpreter (if peeded) | | | /2: | AM/PM |
| Interpreter (if needed) Date | | Time | (CIIC | ie one) |

PLEASE UPLOAD COMPLETED CONSENT FORM TO EPIC.

Revision 2.1 dated: 03-31-2025 Consent document date: 03-31-2025 St. Jude Children's Research Hospital

IRB NUMBER: 22-1021